CLINICAL TRIAL: NCT02689622
Title: Best PREDICTive FactOR of Overall Survival Among Geriatric Assessment Tools and Disease Related Factors in Elderly Patients With High Risk Myelodysplastic Syndromes.
Brief Title: PREDICTive FactOR of Overall Survival Among Geriatric Assessment Tools and Disease Related Factors in Elderly Patients With High Risk Myelodysplastic Syndromes.
Acronym: PREDICTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14 7429 07
Record Dates: First submitted 2015-12-14; First posted 2016-02-24 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: Hematology; Elderly; High Risk Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Physical Functional Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation of disease prognostic factors (Experimental): Research of disease-related factors, research of comorbidities, geriatric assessment (Mini Mental Status Examination (MMSE), Geriatric Depression Scale-15, Mini Nutritional Assessment, Short Physical Performance Battery, grip strength, Fried criteria, Activities of Daily Living (ADL), Instrumental-ADL, G8, self-reported health status, quality of life Quality of Life Questionnaire-C30, Elderly Cancer Patients-14, EQ5D) at inclusion. At 3 months ADL and physical performance. Grade 3/4 toxicities and serious adverse events will be assessed during 6 months after inclusion (using NCI-COMMON TERMINOLOGY CRITERIA version 2.0) whatever treatment type (chemotherapy, supportive care).
  Interventions: Other: research of disease-related factors; Other: research of comorbidities; Other: physical performance

INTERVENTIONS:
Other: research of disease-related factors — included in IPSS and IPSS-R, lactate dehydrogenase, ferritin level, transfusion- dependence, molecular markers as genes mutations
Other: research of comorbidities — HCT-Comorbidity Index, MDS-Comorbidity Index, Adult Comorbidity Evaluation-27, Cumulative Illness Rating Scale-G
Other: physical performance — Activities of Daily Living and physical performance

SUMMARY:
No prospective study was conducted in elderly patients with cancer to assess the relative value of disease-related and patient-related prognosis factors. Patient-related prognostic factors have been highlighted in elderly patients with cancer resulting in the necessity of a geriatric assessment. The impact on overall survival of all of these factors was recognized in elderly people with cancer but remains unknown in High Risk Myelodysplastic Syndromes (HR-MDS). Therefore this information could be crucial to better select geriatric assessment domains relevant for the prediction and to recommend simplified tool after stratification of geriatric assessment domains thanks to their predictive value.

The main hypothesis is that patient-related factors will have a better capacity to predict survival and treatment tolerance than disease-related factors in HR-MDS aged 75 and over and that the predictive value will be different among assessment tools which allows a selection of reduced number of tools for clinical use.

To best knowledge estimation of predictive value of geriatric assessment tools remains unknown and explains why no standardization of practice exists. In testing all tools at the same cohort of patients allows to compare different tools and to define minimal and optimal geriatric assessment for HR-MDS. To determine the best strategy of geriatric assessment will allow in a second time to measure the impact of the use of this geriatric standardized evaluation by comparing patients'care and prognosis according to the use or not by the doctors of the new scores.

Research outcomes are various medical, economic and ethic. Medical because decision-making will be improved with simplified geriatric assessment; economic because a better knowledge of geriatric assessment will improve treatment toxicity prevention and decrease treatment costs. Ethic will be associated with this project because a better knowledge of geriatric assessment tools to predict survival and tolerance treatment could improve the choice of best supportive care if prognosis markers are not favorable to active therapy. This project could induce important modification of practice in this area to an improved personalized treatment and simplification of geriatric assessment allowing a large diffusion in hospitals and clinics.

ELIGIBILITY:
inclusion criteria:

* Diagnosis of HR-MDS inferior to 6 weeks,
* No treatment received before inclusion,
* IPSS superior to 1 (intermediate 2 and high risk IPSS categories),
* Social system affiliation,
* Informed consent signed.

exclusion criteria:

* Patient eligibility to stem cell transplantation,
* IPSS inferior or egal 1 (low or intermediate 1 IPSS),
* Concomitant investigational trial participation, which could interfere,
* Patients under legal protection.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 157 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
IPPS score | 1 year

SECONDARY OUTCOMES:
percentage of patients who had adverse events grade 3 or higher or having a serious adverse event | 6 months
difference of geriatric assessment score between day 1 and 3 month | day 1 and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Odile BEYNE-RAUZY, MD, Principal Investigator — University Hospital, Toulouse
Locations (31):
- France (30):
  - Hôpital Sud, Amiens
  - Chu Angers, Angers
  - CH Annecy, Annecy
  - CH Henri Duffaut, Avignon
  - CH Blois, Blois
  - CH Boulogne sur mer, Boulogne-sur-Mer
  - CH Sud Francillien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHU Albert Michallon, Grenoble
  - CH Versailles, Le Chesnay
  - CH du Mans, Le Mans
  - CH de Lens, Lens
  - Hôpital saint vincent de paul - Institut Catholique, Lille
  - CHU Limoges, Limoges
  - Ch Lyon Sud, Lyon
  - Institut Paoli Calmette, Marseille
  - CH de Meaux, Meaux
  - Chu Brabois, Nancy
  - Chu Hotel Dieu, Nantes
  - Hôpital de l'archet I, Nice
  - Hôpital COCHIN, Paris
  - Hôpital St Louis, Paris
  - CH Saint Jean, Perpignan
  - CHU Poitiers, Poitiers
  - CH René Dubos, Pontoise
  - Hôpital Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - CH St Malo, St-Malo
  - CHU Toulouse, Toulouse
  - Hôpital Bretonneau, Tours
- CH Princesse Grâce, Monaco, Monaco

IPD SHARING:
Plan to Share IPD: No